CLINICAL TRIAL: NCT07061327
Title: Effectiveness of an Online Educational Intervention to Improve Parents' Fever Management Practices: A Randomized Controlled Trial
Brief Title: Online Training to Improve Parents' Fever Management Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Gamzegül ALTAY, Assistant Professor of Child Health and Disease Nursing, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AltayGamzegül
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Fever; Parents
Keywords: Parent, Fever, Management, Online
MeSH Terms: conditions — Fever

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Online fever management training
  Interventions: Behavioral: Online fever management
- Control group (No Intervention): Fever management training will not be provided

INTERVENTIONS:
Behavioral: Online fever management — Online training application will be carried out via Whatsapp
  Arms: Intervention group

SUMMARY:
This study was planned to evaluate the effects of education provided to parents via WhatsApp on fever management. This research is a randomized controlled trial. The study includes parents who were reached via social media between April 2025 and July 2025 and who agreed to participate in the study voluntarily. The research sample will consist of mothers reached on the specified dates. The "Sociodemographic Data Collection Form", "Fever Management Questionnaire", "Fever Management Scale" and "E-Health Literacy" scale will be used to collect data.

DETAILED DESCRIPTION:
Type of Research: The research was planned as a single-blind, randomized controlled experimental design to evaluate the effect of education provided to parents via WhatsApp on parents' fever management.

Place and Time of the Research: The research will be conducted between April 2025 and July 2025 with parents who were reached via social media and agreed to participate in the study voluntarily.

Research Universe and Sample: The study sample consists of parents with children aged 0-5. The sample size of the research was calculated using the G*Power 3.1.9.7 program. In the calculation, the sample calculation was made for the Two-Way Mixed Design ANOVA analysis, considering the 2-group (Experimental Group, Control Group) and 3-measurement (Pretest, Posttest, Permanence test) research design. In the calculation, the effect size was calculated as 0.15 (f = 0.15), 5% margin of error (α = 0.05) and 80% power (1-β = 0.80) and the sample size for each group was calculated as 37. Considering the possibility of data loss, the sample size for each group was increased by 10%. As a result, it was planned to include 41 patients in each group and a total of 82 patients in the sample (Cohen, 1988; Faul, 2007). Only one parent from each family will be included in the study. Sample selection will be made using stratified randomization and random sampling methods. This method ensures homogeneous distribution between the groups. When creating the intervention and control groups, stratification will be made by targeting the age of the children and the educational status of the parents. The distribution of the parents to the intervention and control groups will be done randomly.

Intervention The training modules to be prepared by the researchers in line with current guidelines and literature will be sent via WhatsApp in the form of written text or audio recording. The training will last for 6 weeks and information will be provided about the content of the prepared training module every week and parents' questions will be answered. During the training, the "Fever Management Skills for Parents" guide, which will be created by the researchers after receiving expert opinion, will be given by the researchers in WhatsApp groups. This training module is planned to consist of 6 sub-modules (Definition and importance of fever, fever measurement, fever-reducing interventions, fluid intake and nutrition in children with fever, when to apply to a health institution, strategies to reduce fear of fever). Each module includes information on fever management for parents at home. The content of the training will be shared in groups as text and audio recordings. Each audio recording message will last approximately 5 to 10 minutes.

Data Collection The researchers will provide preliminary information about the study to the parents who agree to participate in the study and collect data after obtaining their digital consent. In the data collection process, pre-test and post-test data will be collected online.

Control group: At the end of the study, training materials prepared on fever management based on the "Equality Principle" will be shared with the parents in the control group.

Intervention group: Before the training modules to be prepared by the researchers are sent to the parents in the intervention group, the pre-test data of the Sociodemographic Data Collection Form, Fever Management Survey, and E-Health Literacy Scale will be collected online. After the pre-test data is collected, the training content prepared as 6 modules will be shared as one module every week and the parents' questions will be answered. Post-test data will be collected at the end of the training.

Ethical Principles of the Study Ethical approval (Issue No: E-40465587-050.01.04-1412, Decision No: 2025/92) was obtained from the Ethics Committee of the Recep Tayyip Erdoğan University Faculty of Medicine in order to conduct the study. The purpose of the study was explained to the parents who met the research group criteria, the questions asked were answered, and their verbal and written consents were obtained. The parents were informed that the data collected during the study would be processed confidentially and anonymously, would not be used outside the study in question, and that they could withdraw from the study at any time. Since the study was based on the use of data obtained from people and therefore due to the necessity of protecting personal rights, the relevant ethical principles of "Informed Consent", "Voluntariness" and "Protection of Confidentiality" were followed. After the data collection process was completed with the mothers in the control group, the training modules were shared and the "Equality Principle" was tried to be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Being a mother
* Having a child between the ages of 0-5
* Agreeing to participate in the research voluntarily
* Not having any chronic diseases in the child
* Not having any chronic diseases

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Fever management survey | 3 month
  The fever management survey was created by the researchers by reviewing the relevant literature and examining the institutional guidelines (Sullivan and Farrar, 2011; El-Radhi, 2012; Yalnızoğlu Çaka et al., 2015; Chiappini et al., 2017; Elkon-Tamir et al., 2017; Kelly et al., 2019; Green et al., 2021; NICE, 2021; Vicens-Blanes et al., 2023). The survey form contains a total of 28 questions evaluating fever in children, fever detection, fever management and antipyretic use. Each question was prepared according to the 5-point Likert type (1 = I completely disagree - 5 = I completely agree). The participant can get a minimum of 28 and a maximum of 140 points from the survey. As the score obtained from the survey increases, the level of correct fever management in children by the parents also increases. Expert opinions were received from 7 faculty members working in the field of child health and disease nursing for the survey. Experts gave 1-4 points to each question (1=A lot of change is
E-health literacy scale | 3 month
  The scale developed by Norman and Skinner (2006) was adapted to Turkish by Tamer Gencer (2017). The scale, consisting of 8 items, was designed as a 5-point Likert scale as follows: 1=I completely disagree, 2=I disagree, 3=I am undecided, 4=I agree, 5=I completely agree. The lowest score from the scale is 8, and the highest score is 40. As the score from the scale increases, the level of e-health literacy increases. The Cronbach Alpha value of the scale is 0.86. In order to use the scale in the study, permission to use the scale was obtained from the researcher who adapted the scale to Turkish (Tamer Gencer, 2017).
Parental Fever Management Scale | 3 month
  The scale, developed by Walsh and Edwards in 2008 to assess fever management in parents, was adapted to Turkish by Çınar et al. (22) in 2013. The scale consists of eight questions. The questions are usually asked to question what parents do when their child has a fever. Participants can choose answers to Likert-type questions rated as "(1) never, (2) rarely, (3) sometimes, (4) often, (5) always". The lowest score on this scale can be 8 and the highest score can be 40. Higher scores indicate more fever management practices, while lower scores indicate less fever management practices. The Cronbach Alpha reliability coefficient of the scale is 0.79.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The aim is to share the research after it is published.

REFERENCES:
- [Derived] Altay G, Karaaslan MM, Celik I. The effectiveness of a WhatsApp-based educational intervention aimed at improving mothers' fever management: A randomized controlled trial. J Pediatr Nurs. 2026 Jan 14;87:146-153. doi: 10.1016/j.pedn.2026.01.013. Online ahead of print. PMID 41539254